CLINICAL TRIAL: NCT07232381
Title: Turkish Validity and Reliability Study of Diabetes-Specific Nutrition Knowledge Questionnaire in Adolescents With Type 1 Diabetes
Status: Completed | Type: Observational
Sponsor: Yasemin Atik Altinok (Other)
Collaborators: Izmir Tinaztepe University (Other)
Responsible Party: Sponsor-Investigator, Yasemin Atik Altinok, Dr.Dyt., Ege University
Organization: Ege University (Other)
Other Study IDs: 23-11.1T/35
Record Dates: First submitted 2025-05-27; First posted 2025-11-18 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 3 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Child: The population of the study consists of adolescent individuals with type 1 diabetes between the ages of 10 and 19 who were diagnosed with diabetes at least one year ago. The sample of the study consists of adolescents with type 1 diabetes and their parents, who were followed up for diabetes at Ege University Faculty of Medicine Department of Child Health and Diseases, Pediatric Endocrine Department in Izmir, who met the inclusion criteria for the study and approved the informed consent form.
- Parent: The population of the study consists of adolescent individuals with type 1 diabetes between the ages of 10 and 19 who were diagnosed with diabetes at least one year ago. The sample of the study consists of adolescents with type 1 diabetes and their parents, who were followed up for diabetes at Ege University Faculty of Medicine Department of Child Health and Diseases, Pediatric Endocrine Department in Izmir, who met the inclusion criteria for the study and approved the informed consent form.

SUMMARY:
It is aimed to contribute to the Turkish Nutrition Sciences literature and shed light on the studies of future generations by establishing the Turkish validity and reliability of this scale, which was developed for adolescents with type 1 diabetes and their parents and was designed to evaluate general and diabetes-specific nutrition knowledge.

Hypotheses:

* H1: Diabetes-Specific Nutrition Information Scale for Adolescents with Type 1 Diabetes is a reliable tool for the Turkish population.
* H2: Diabetes-Specific Nutrition Information Scale for Adolescents with Type 1 Diabetes is a valid tool for the Turkish society.
* H3: Individuals with higher scores on the Diabetes-Specific Nutrition Information Scale in Adolescents with Type 1 Diabetes have better metabolic control.
* H4: Diet quality of individuals with higher scores on the Diabetes-Specific Nutrition Information Scale for Adolescents with Type 1 Diabetes is better.

DETAILED DESCRIPTION:
The aim is to analyze the validity and reliability of the Diabetes-Specific Nutrition Information Scale in Adolescents with Type 1 Diabetes for the Turkish population. In this context, the relationship between nutritional knowledge levels, glycemic control and diet quality will be investigated with the Nutrition Knowledge Scale in Adolescents with Type 1 Diabetes.

The sample of the study consists of individuals between the ages of 10-19 with Type 1 diabetes registered at Ege University Faculty of Medicine, Department of Child Health and Diseases, Pediatric Endocrine Department, in Izmir province, and their parents. In the first stage, it will be validated with the Brislin method for Turkish language validity. Later, validity and reliability analysis will be conducted. The relationship between individuals' nutritional knowledge levels and diet quality (adapted to Healthy Eating Index-2015 TÜBER-2022) and metabolic control (with last measured HbA1c) will be examined. The case report form created for this purpose, the food consumption monitoring form, SYI-2015 adapted to TÜBER 2022 and the Turkish version of the Diabetes-Specific Nutrition Information Scale in Adolescents with Type 1 Diabetes will be used.

ELIGIBILITY:
Inclusion Criteria:

* duration of T1D of at least one year,
* regular follow-up of at least 1 year,
* no major medical problems (celiac disease, cystic fibrosis, psychiatric disorders, and communication difficulties)
* the insulin requirement was > 0.5 IU/kg/day

Exclusion Criteria:

* type 1 diabetes duration less than 1 year
* no regular follow-up of at least 1 year
* have major medical problems (celiac disease, cystic fibrosis, psychiatric disorders, and communication difficulties) the requirement was <0.5 IU/kg/day

Ages: 9 Years to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: adolescents witt type 1 diabetes
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-03-30 (Actual); Study Completion 2024-07-10 (Actual)

PRIMARY OUTCOMES:
Nutritional Knowledge | 3 day
  If your nutritional knowledge score is high your diet is healthy.

CONTACTS AND LOCATIONS:
Locations (1):
- Ege University, Medical Faculty, Division of Pediatric Endocrinology, Izmir, İzmir, Turkey (Türkiye)